CLINICAL TRIAL: NCT02013154
Title: A Multi-part, Phase 1, Multi-center, Open-label Study of DKN-01 as a Monotherapy or in Combination With Paclitaxel or Pembrolizumab in Patients With Relapsed or Refractory Esophagogastric Malignancies
Brief Title: A Study of DKN-01 in Combination With Paclitaxel or Pembrolizumab
Acronym: P102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P102; DKN-01; LY2812176; KEYNOTE-731 (Other: Merck)
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Neoplasms; Adenocarcinoma of the Gastroesophageal Junction; Gastroesophageal Cancer; Squamous Cell Carcinoma; Gastric Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell | interventions — Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- DKN-01 150 mg plus paclitaxel (Experimental): DKN-01 150 mg administered on Days 1 and 15 and paclitaxel 80 mg per meter squared of body surface area (mg/m2) administered on Days 1, 8, 15, and 22
  Interventions: Drug: DKN-01 150 mg; Drug: Paclitaxel
- DKN-01 300 mg plus paclitaxel (Experimental): DKN-01 300 mg administered on Days 1 and 15 and paclitaxel 80 mg per meter squared of body surface area (mg/m2) administered on Days 1, 8, 15, and 22
  Interventions: Drug: Paclitaxel; Drug: DKN-01 300 mg
- DKN-01 150 mg plus pembrolizumab (Experimental): DKN-01 150 mg administered on Days 1 and 15 and pembrolizumab 200 mg administered on Day 1
  Interventions: Drug: DKN-01 150 mg; Drug: Pembrolizumab
- DKN-01 300 mg plus pembrolizumab (Experimental): DKN-01 300 mg administered on Days 1 and 15 and pembrolizumab 200 mg administered on Day 1
  Interventions: Drug: Pembrolizumab; Drug: DKN-01 300 mg
- DKN-01 300 mg monotherapy (Experimental): DKN-01 300 mg administered on Days 1 and 15
  Interventions: Drug: DKN-01 300 mg

INTERVENTIONS:
Drug: DKN-01 150 mg — Administered by IV infusion
  Arms: DKN-01 150 mg plus paclitaxel; DKN-01 150 mg plus pembrolizumab
Drug: Paclitaxel — Administered by IV infusion
  Other Names: Taxol
  Arms: DKN-01 150 mg plus paclitaxel; DKN-01 300 mg plus paclitaxel
Drug: Pembrolizumab — Administered by IV infusion
  Other Names: Keytruda
  Arms: DKN-01 150 mg plus pembrolizumab; DKN-01 300 mg plus pembrolizumab
Drug: DKN-01 300 mg — Administered by IV infusion
  Arms: DKN-01 300 mg monotherapy; DKN-01 300 mg plus paclitaxel; DKN-01 300 mg plus pembrolizumab

SUMMARY:
A study to evaluate the safety and tolerability of DKN-01 in combination with weekly paclitaxel or pembrolizumab in participants with relapsed or refractory Esophagogastric Malignancies

DETAILED DESCRIPTION:
This is a dose-escalating, open-label study conducted in multiple parts (Part A dose-escalation, Parts B-F expansion cohorts, and a monotherapy substudy). Parts A-E (DKN-01 plus paclitaxel) and the DKN-01 monotherapy substudy includes 28-day cycle treatment cycles; Part F (DKN-01 plus pembrolizumab) includes 21-day treatment cycles. Depending on their cancer type, subjects with histologically confirmed recurrent or refractory esophageal, gastro-esophageal junction tumors, or gastric adenocarcinoma will be enrolled in each study part to receive DKN-01 150 mg or 300 mg in combination with paclitaxel or pembrolizumab. Subjects who are unable to receive paclitaxel or pembrolizumab for any reason are allowed to receive single agent DKN-01 300 mg as part of a monotherapy substudy. Results are reported by treatment group, irrespective of the study part in which the subject was enrolled.

ELIGIBILITY:
Inclusion Criteria:

In advanced esophagogastric malignancies:

* Participants with histologically confirmed recurrent or metastatic esophageal or gastro-esophageal junction squamous cell or adenocarcinoma or gastric adenocarcinoma with Wnt Signaling Alterations
* Participants must be refractory or intolerant to at least one prior therapy(ies) for metastatic or locally advanced disease

  * If prior therapy consisted of palliative chemoradiation therapy, it will be considered one line of therapy
  * Prior treatment with paclitaxel as part of a definitive therapy regimen is acceptable. Patients who are unable to receive paclitaxel for any reason will be allowed to receive DKN-01 as a single agent.
  * Prior treatment anti- programmed death-1 (PD-1)/ anti-PD-ligand 1 (PD-L1) monoclonal antibody (mAb) is permitted in patients provided the patient's disease is primary refractory, and the patient is not intolerant of pembrolizumab. Patients who are not eligible to receive pembrolizumab will be allowed to receive single agent DKN-01
* Tumor tissue for mandatory evaluation
* Must have one or more tumors measurable on radiographic imaging as defined by the Response Evaluation Criteria in Solid Tumors (RECIST). Patients with evaluable but not measurable disease per RECIST criteria may be enrolled with the approval of the medical monitor.
* Must be ≥18 years of age
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale. A performance status of 2 on the ECOG scale may be entered upon the review and approval of the medical monitor
* Disease-free of active second/secondary or prior malignancies for equal to or over 2 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast
* Acceptable liver, renal, hematologic and coagulation function
* For men and women of child-producing potential, the use of effective contraceptive methods during the study and for 6 months following the last dose of study drug

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia
* Fridericia-corrected QT interval (QTcF) > 470 msec (female) or > 450 (male), or history of congenital long QT syndrome.
* Active, uncontrolled bacterial, viral, or fungal infections, within 7 days of study entry requiring systemic therapy
* Known to be human immunodeficiency virus (HIV) positive, have hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb) unless HCV RNA is undetected/negative.
* Serious nonmalignant disease
* Pregnant or nursing women
* History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on MRI scan that are symptomatic and clinically significant.
* Systemic central nervous system (CNS) malignancy or metastasis.
* Clinically significant peripheral neuropathy at the time of study entry. Patients with pre-existing peripheral neuropathy will be allowed to receive single agent DKN-01
* Known osteoblastic bony metastasis
* History of known or suspected autoimmune disease with the specific exceptions of vitiligo, atopic dermatitis, or psoriasis not requiring systemic treatment.
* Clinically-significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis.
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Treatment with surgery or chemotherapy within 21 days prior to study entry (42 days for nitrosoureas or mitomycin C)
* Treatment with low dose chemotherapy concurrent with radiation within 14 days prior to study entry
* Treatment with radiation therapy within 14 days prior to study entry
* Treatment with any other investigational agent within 30 days prior to study entry
* Previously treated with an anti-DKK-1 therapy
* Participants who have a history of hypersensitivity reactions to TAXOL® or other drugs formulated in Cremophor® EL (polyoxyethylated castor oil). Patients who exhibit these hypersensitivities will be eligible to receive single agent DKN-01.
* Significant allergy to a pharmaceutical therapy that, in the opinion of the investigator, poses an increased risk to the participant
* Treatment with corticosteroids (≥ 10 mg per day prednisone or equivalent) or other immune suppressive drugs within the 14 days prior to study entry
* Active substance abuse
* Receipt of any live vaccines within 30 days before the first dose of study treatment and while participating in the study
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* History of interstitial lung disease
* Intolerance or severe hypersensitivity (≥Grade 3) to pembrolizumab and/or of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose limiting toxicities in each treatment arm | Baseline to End of Cycle 1 (each cycle is 28 days, except each cycle is 21 days when DKN-01 is administered with pembrolizumab)
Number of subjects with treatment emergent adverse events related to study treatment (DKN-01 as monotherapy or in combination with paclitaxel or pembrolizumab) | Baseline until 30 days after last dose of study drug

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (approximately 3 months)
Duration of Response (DoR) | Baseline to study completion (approximately 3 months)
Overall Survival (OS) | Baseline to study completion (approximately 3 months)
Progression Free Survival (PFS) | Baseline to study completion (approximately 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndi Sirard, MD, Study Director — Leap Therapeutics, Inc.
Locations (10):
- United States (10):
  - Cedars Sinai Medical Care Foundation, Los Angeles, California
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Tennessee Oncology / Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University / VICC, Nashville, Tennessee
  - Mary Crowley Cancer Center, Dallas, Texas
  - CTRC @ The University of Texas Health Science Center at San Antonio, San Antonio, Texas